CLINICAL TRIAL: NCT06979856
Title: Short, Animated Storytelling Videos to Reduce Smartphone Addiction in the US: Protocol for an Online, Randomized Controlled Trial
Brief Title: Short, Animated Storytelling (SAS) Videos to Reduce Smartphone Addiction in the US
Acronym: SAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Maya Adam, Clinical Associate Professor of Pediatrics, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 80171
Record Dates: First submitted 2025-05-06; First posted 2025-05-20 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Smartphone Addiction
Keywords: Addictive Behavior; Smartphone addiction; screen time; digital well-being; mental health
MeSH Terms: conditions — Internet Addiction Disorder; Behavior, Addictive; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Animated videos (Experimental): Participants will watch two short, animated storytelling videos about digital addiction.
  Interventions: Behavioral: Short animated videos
- Informational Control (Active Comparator): Participants will read a fact sheet containing written information and statistics about smartphone usage.
  Interventions: Behavioral: Informational Control
- Do-nothing control (No Intervention): Participants will only complete the surveys. Participants do not receive any intervention or information about digital addiction.

INTERVENTIONS:
Behavioral: Short animated videos — The short animated videos (approximately 2 minutes each) draw attention to the dangers of smartphone addiction.
  Arms: Animated videos
Behavioral: Informational Control — A short fact sheet presenting written information and statistics about smartphone usage.
  Arms: Informational Control

SUMMARY:
This study will test the effect of exposure to short, animated storytelling videos on participants' perceived risk of smartphone overuse immediately after exposure, two weeks later and four weeks later.

ELIGIBILITY:
Inclusion Criteria:

* English Speaking
* Own a Smartphone
* Live in the US

Exclusion Criteria:

* None

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6000 (Estimated)
Dates: Start 2026-02-09 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Smartphone Addiction Scale (SmAS) score | Baseline, 2 weeks and 4 weeks post intervention
  SmAS is a short 10 item validated scale measuring smartphone addiction. The minimum value is 10 and the maximum value is 60 for this scale.
Mobile Phone Attachment Scale - Anxious Attachment Sub Scale (MPAS-AA) | Baseline, immediate post-intervention (up to 24 hours), 2 weeks and 4 weeks post intervention
  The MPAS Anxious Attachment subscale comprises 7 items rated 1 (not at all true) to 5 (extremely true). Subscale scores were computed as the mean of the 7 items (range 1-5), with higher scores indicating greater anxious attachment to one's mobile phone. The MPAS-AA has demonstrated good internal consistency (α=.87) and external validity.

SECONDARY OUTCOMES:
Mobile Phone Attachment Scale - Addiction Sub Scale (MPAS_Addiction) | Baseline, 2 weeks and 4 weeks post intervention
  Mobile phone addiction will be assessed with the MPAS Addiction subscale (6 items). Items are rated on a 5-point scale from 1 = not at all true to 5 = extremely true; responses are averaged to create a subscale score (range 1-5), with higher scores indicating greater addictive/problematic mobile phone use.
Perceived Danger of Smartphone Overuse measured using a visual analogue scale (VAS) | Baseline, immediately post intervention exposure (up to 24 hours), 2 weeks and 4 weeks post intervention exposure
  Perceived danger of smartphone overuse will be assessed with a single-item 10-point slider (visual analogue-type scale) ranging from 0 = not at all dangerous to 10 = extremely dangerous. Higher scores indicate greater perceived danger.
Self-reported daily smartphone use (past 2 weeks) | Baseline, 2 weeks and 4 weeks post intervention exposure
  Self-reported daily smartphone use will be assessed via a single self-report item asking participants: 'On average, how many hours per day did you use your phone over the past two weeks?' Responses are recorded in 6 ordered categories: <1 h, 1-2 h, 2-4 h, 4-6 h, 6-8 h, >8 h, with higher categories indicating greater daily use.
Self-perceived smartphone addiction (single item; Olsen) | Baseline, immediately post intervention exposure (up to 24 hours) 2 weeks and 4 weeks post intervention exposure
  Self-perceived smartphone addiction will be assessed using Olsen's single-item smartphone addiction measure, asking agreement with the statement 'I am addicted to my smartphone' on a 6-point Likert scale from Strongly disagree (1) to Strongly agree (6). Higher scores indicate greater self-perceived smartphone addiction.

CONTACTS AND LOCATIONS:
Overall Officials: Maya U Adam, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No